CLINICAL TRIAL: NCT05697874
Title: International Rare Brain Tumor Registry
Acronym: IRBTR
Status: Recruiting | Type: Observational
Sponsor: Children's National Research Institute (Other)
Responsible Party: Principal Investigator, Adriana Fonseca, Oncologist, Children's National Research Institute
Other Study IDs: STUDY00000324
Record Dates: First submitted 2023-01-23; First posted 2023-01-26 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Astroblastoma; BCOR ITD Sarcoma; CNS Sarcoma; Unclassified Tumor, Malignant
Keywords: Rare Brain Tumor; Pediatric Brain Tumor Registry; Unclassifiable tumor; Pediatric Neuro-Oncology; Rare Disease
MeSH Terms: conditions — Neoplasms, Neuroepithelial; Neoplasms; Rare Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Tumor tissue, blood, urine, cerebrospinal fluid (CSF). Samples are collected only if part of a clinically indicated procedure from enrolled individuals.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- CNS Sarcoma: Patients diagnosed with Central nervous system (CNS) sarcomas
- BCOR-altered: Patients diagnosed with tumors characterized by alterations in the BCOR gene.
- Astroblastoma/MN-1- altered: Patients diagnosed with Astroblastomas/MN-1 alterations
- Unclassifiable tumors: Patients diagnosed with histologically ambiguous tumors or tumors that fail to classify with the current diagnostic methods.
- Other Rare Brain tumors: Patients diagnosed with other rare brain tumors that do not meet the criteria for cohorts 1-4.

SUMMARY:
The objective of the International Rare Brain Tumor Registry (IRBTR) is to better understand rare brain tumors through the collection of biospecimens and matched clinical data of children, adolescents, and young adult patients diagnosed with rare brain tumors.

DETAILED DESCRIPTION:
The International Rare Brain Tumor Registry (IRBTR) is a prospective observational study that will collect tumor samples and matched clinical and radiological data to better understand the outcomes of patients with rare brain tumors in particular: CNS sarcoma, BCOR, MN-1 altered tumors, PLAG/L1, and other rare or unclassified rare brain tumors.

Data collected include demographics, disease characteristics, treatment information, radiological imaging, and biospecimen collection if available ( tumor tissues Patients will be followed longitudinally to obtain outcome data. Data collection will continue for approximately 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a known or suspected CNS Sarcoma.
* Patients with a known or suspected BCOR-altered brain tumor
* Patients with a known or suspected Astroblastoma/NM-1 altered brain tumor
* Patients with known or suspected histologically ambiguous/unclassifiable brain tumor
* Patients with a known or suspected rare brain tumor.
* Signed informed consent by patient/ parent or guardian (assent where applicable) to participate in the study.

Exclusion Criteria:

* The patient has an extra-CNS primary tumor.
* The patient is older than 46 years of age at diagnosis.
* The patient or family is not willing to participate or does not sign informed consent.

Max Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population will include patients who have completed the informed consent process and are <= to 45 years of age at diagnosis of the following: CNS Sarcoma, BCOR-altered tumor, Astroblastoma/MNI-1 altered tumors, histologically ambiguous/unclassifiable brain tumor, rare brain tumor. Patients from anywhere in the world are eligible for enrollment.
Sampling Method: Non-Probability Sample
Enrollment: 5800 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2033-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Event-free Survival | 10 years
  The primary outcome measure will be time from diagnosis to an event, defined as the occurrence of progression or recurrence of the disease, occurrence of a second malignant neoplasm, or death from any cause. Each cohort will be analyzed separately.

SECONDARY OUTCOMES:
Molecular characterization | 10 years
  To determine molecular characteristics of each cohort using somatic and germline SNV calling, methylation profiling, fusion calling and gene expression profiling. Molecular findings will be correlated with clinical characteristics to identify risk factors and subgroup-specific therapeutic susceptibilities.
Radiological characterization | 10 years
  To analyze conventional and advanced imaging findings (including diffusion weighted imaging) of each cohort and correlate them with clinical, histopathology and molecular data (radiogenomics).

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Fonseca, MD, Principal Investigator — afonsecash@childrensnational.org
Locations (4):
- United States (4):
  - Nathan Robison, Los Angeles, California
  - Marie Jaeger-Krause, San Francisco, California
  - Children's National Hospital, Washington D.C., District of Columbia
  - Scott Raskin, Cincinnati, Ohio

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared with other researchers.